CLINICAL TRIAL: NCT07203066
Title: Effects of Oxaliplatin-Induced Peripheral Neuropathy on Hand Function, Grip Strength and Quality of Life in Colorectal Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Fenerbahce University (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Principal Investigator, Ozge Koseoglu, research assisstant, Fenerbahce University
Other Study IDs: TY-2025-2260
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy; Oxaliplatin Induced Peripheral Neuropathy in Cancer Patients; Hand Strength
Keywords: Colorectal Cancer; Oxaliplatin; Chemotherapy-Induced Peripheral Neuropathy; Hand Function
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational only — observational only

SUMMARY:
The aim of this study is to investigate the effects of oxaliplatin-induced peripheral neuropathy on hand function, grip strength, and quality of life in colorectal cancer patients. Assessing the motor symptoms of CIPN and sharing the results in clinical settings will help guide evidence-based practices and interventions.

DETAILED DESCRIPTION:
Oxaliplatin is a chemotherapy drug frequently used in the treatment of colorectal cancers, the third most common type of cancer. However, oxaliplatin is associated with long-term neurotoxicity, the most common dose-limiting side effect. Chemotherapy-induced peripheral neuropathy (CIPN) is a common adverse effect of platinum-based chemotherapy agents, such as oxaliplatin. CIPN limits patients' ability to tolerate treatment and adversely affects long-term quality of life and physical functionality. In individuals undergoing colorectal cancer treatment, the prevalence of CIPN has been reported as 58% at 6 months, 45% at 12 months, 32% at 24 months, and 24% at 36 months post-treatment. Additionally, oxaliplatin exhibits a "coasting phenomenon," in which CIPN symptoms continue to worsen for approximately 3 months after treatment. Although the incidence and sensory symptoms of oxaliplatin-induced CIPN during chemotherapy have been well documented, the chronic-phase motor symptom burden of oxaliplatin-induced CIPN has not been reported. Studies investigating the motor aspects of CIPN are insufficient, and further research is needed to determine its prevalence, progression, and impact on functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemotherapy due to a diagnosis of locally advanced or metastatic colorectal cancer,
* Having received at least 3 cycles of single or combined oxaliplatin-based chemotherapy,
* Aged 20 years or older,
* No speech or hearing impairments,
* Voluntary participation in the study.

Exclusion Criteria:

* Development of peripheral neuropathy due to causes other than chemotherapy (e.g., tumor compression, nutritional disorders, infections, or major systemic diseases such as diabetes mellitus),
* Presence of mental or cooperation problems.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer patients who received oxaliplatin based chemotherapy
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-09-24 (Estimated); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength Assessment | baseline only
  Participants' hand grip strength will be evaluated using the Saehan Hydraulic Hand Dynamometer (SAEHAN Corporation, Yangdeok-Dong, Masan, South Korea) to assess the functional status of the upper extremity and clinical outcomes.
Finger Grip Strengths (Tip, Key, and Palmar Grip) | baseline only
  A hydraulic pinch gauge will be used to measure finger grip strengths.
Hand Function Assessment (Duruöz Hand Index) | baseline
  Hand function related to daily activities will be assessed using the Duruöz Hand Index questionnaire. This questionnaire consists of 18 items covering five domains: kitchen tasks, dressing, personal hygiene, work activities, and other activities. Each item is scored on a scale from 0 to 5.
Hand Function Assessment (Michigan Hand Outcomes Questionnaire) | baseline
  Overall hand function, including parameters such as pain, aesthetic perception, and patient satisfaction, will be assessed using the Michigan Hand Outcomes Questionnaire (MHQ). The MHQ was developed in 1998 by hand surgeon Chung and colleagues Pillsbury, Walters, Hayward, and Arbor. The questionnaire consists of six domains: overall hand function, activities of daily living, work performance, pain, aesthetics, and patient-reported hand function. Scores range from 0 to 100. Responses are rated on a scale of 1 to 5 and then normalized to obtain scores for each subdomain.
Fine Motor Skill Assessment (Minnesota Manual Dexterity Test) | baseline
  Fine motor skills will be assessed using the Minnesota Manual Dexterity Test (MMDT), which evaluates unilateral and bilateral manual performance of the upper extremities through placement and turning tasks. In the placement test, participants are required to place 60 cylinders one by one into holes on a board as quickly as possible using one hand. The dominant and non-dominant hands are evaluated separately. In the turning test, at the start of the test, all 60 cylinders are placed in the holes. Participants are asked to pick up each cylinder with one hand, rotate it, and return it to the hole using the other hand, repeating this process for all 60 cylinders individually.
Nine-Hole Peg Test (NHPT) | Baseline
  The Nine-Hole Peg Test is a standardized, well-established, and reliable tool for assessing hand function.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | baseline
  Developed in 1987, the EORTC QLQ-C30 is the most widely used quality of life questionnaire in cancer research and clinical practice. It consists of three subdimensions: overall well-being, functional performance, and symptoms. The questionnaire includes five functional scales (physical, social, role, emotional, and cognitive functioning), nine symptom scales (fatigue, pain, nausea/vomiting, dyspnea, sleep disturbances, appetite loss, diarrhea, constipation, and financial difficulties), and a global health status scale, totaling 30 items.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) | baseline
  The EORTC QLQ-CIPN20 is a 20-item quality of life questionnaire designed to assess symptoms and impairments related to sensory, motor, and autonomic neuropathy. It has been widely used in oncology studies. Each item is rated on a 4-point scale, and the questionnaire has been validated for clinical and research use.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kannarkat G, Lasher EE, Schiff D. Neurologic complications of chemotherapy agents. Curr Opin Neurol. 2007 Dec;20(6):719-25. doi: 10.1097/WCO.0b013e3282f1a06e. PMID 17992096
- [Background] Wild CP, Weiderpass E, Stewart BW, editors. World Cancer Report: Cancer research for cancer prevention. Lyon (FR): International Agency for Research on Cancer; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK606505/ PMID 39432694